CLINICAL TRIAL: NCT06988527
Title: Treatment Outcomes and Patient Satisfaction of Oral Lichen Planus Treatment
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dar Al Uloom University (Other)
Responsible Party: Principal Investigator, Sally Abd-ElMeniem ElHaddad, Assist. Prof. Oral Medicine and Periodontology, Dar Al Uloom University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 010-012-2022
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-09

CONDITIONS: Erosive Oral Lichen Planus; Atrophic Lichen Planus
MeSH Terms: interventions — Honey; Triamcinolone Acetonide; Ointments

STUDY DESIGN:
Intervention Model Description: * Zα/2=1.96=1.96 (for 95% confidence)
  * Zβ=1.28 (to 90% power)
  * SD=196
  * Δ=1.33
  N≈55.65 N=56
  56 patients diagnosed with Oral Lichen Planus, randomly assigned to one of the 2 groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This was a double-blind, parallel-group clinical trial. Both participants and outcome assessors were blinded to the intervention. The honey in orabase and triamcinolone formulations were prepared to appear similar in color, texture, and packaging to ensure concealment. Identical containers were used for both treatments, and labeling was done using coded identifiers maintained by a third party not involved in the assessment or data analysis. Participants were instructed to apply the provided formulation as directed without being informed of the specific treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I with OLP at buccal mucosa (Experimental): The trial Group (I) (honey in orabase 1: 1 paste), four times daily after meals or rinsing
  Interventions: Drug: Honey in orabase 1: 1 paste
- Group II with OLP at buccal mucosa (Active Comparator): Group (II): triamcinolone acetonide 0.1% ointment, four times daily after meals or rinsing
  Interventions: Drug: Honey in orabase 1: 1 paste

INTERVENTIONS:
Drug: Honey in orabase 1: 1 paste — The experimental drug was manufactured and packed at the Faculty of Pharmacy, Price Sattam University, SA. Production of a mucoadhesive paste involves a step-by-step process. in the final step, honey, comprising 50% of the total composition was thoroughly blended with the prepared base to ensure homogeneity
  Other Names: Triamcinolone acetonide 0.1% ointment

SUMMARY:
The goal of this clinical trial is to assess Honey in orabase (1:1) for treating patients with OLP and improving their quality of life:

The research question aims to answer:

Does honey in orabase (1:1) improve or reduce OLP symptoms compared to the standardized treatment by triamcinolone acetonide 0.1% drug and improve the patient's quality of life?

Participants will:

Take drug ABC or a placebo every day for 4 months Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms and the number of times they use a rescue inhaler

DETAILED DESCRIPTION:
The study comprised 56 patients diagnosed with Oral Lichen Planus, who were randomly selected according to inclusion and exclusion criteria. The subjects were between 35 and 60 years old, capable of complying with the study procedure, and provided informed consent. Exclusion criteria encompassed those with alternative oral mucosal illnesses, systemic problems influencing OLP or wound healing, allergies or sensitivities to honey or triamcinolone, or those receiving systemic corticosteroids or immunosuppressive drugs. Individuals who were pregnant or lactating, as well as those unable to provide informed written consent, were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of oral lichen planus
* Symptomatic OLP lesions (erosive/atrophic)
* Participants are between 35 and 60 years old, who are able to adhere to the study protocol, and sign informed consent.

Exclusion Criteria:

* Patients with other oral mucosal disorders, or systemic conditions influencing OLP or wound healing, allergies or hypersensitivity to honey or triamcinolone
* Patients who administer systemic corticosteroids or immunosuppressive agents.
* Pregnancy or lactation
* Inability to comprehend or adhere to study directives
* Patients who are not able to sign an informed written consent

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment of OLP lesions using OLP score | baseline to 1 year
  will be assessed by OLP score: Thongprasom et al.: score 0 (no lesions), score 1 (mild white striae only with no erythematous areas), score 2 (white striae exhibiting an atrophic area < 1 cm2), score 3 (white striae alongside an atrophic area ≥ 1 cm2), score 4 (white striae in an erosive area < 1 cm2), and score 5 (white striae alongside an erosive area ≥1 cm2). Atrophic OLP was defined as thinning of the oral mucosa, with a smooth red appearance, while erosive OLP involved ulceration and erosion of the mucosal surface.
Pain assessment using Visual analogue scale (VAS) | baseline- to 1 year
  (VAS) is a self-reported score typically consisting of a 10 cm horizontal line from right (best) to left (worst) with verbal descriptions (word anchors: 0 cm: No pain; 1 cm: Hardly notice pain; 2 cm: Notice pain does not interfere with activities; 3 cm: Sometimes distracts me; 4 cm: Distracts me, can do usual activities; 5 cm: Interrupts some activities; 6 cm: Hard to ignore, avoid usual activities; 7 cm: focus of attention, prevent doing daily activities; 8 cm: Awful, hard to do anything; 9 cm: Can not bear the pain, unable to do anything; 10 cm: As bad as it could be, nothing else matters)

SECONDARY OUTCOMES:
Long-term satisfaction of patients with OLP treated with honey, recurrence rates, and quality of life after one year of treatment | baseline to 1 year
  Patient Satisfaction: Measured using a Likert scale questionnaire (e.g., 1-5, where 1 = very dissatisfied and 5 = very satisfied).
  Recurrence % or Complications
  Quality of Life: Reassess by using OHIP-14 at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Sally A ElHaddad, Assist. Prof, Principal Investigator — Dar AlUloom University, SA
Locations (1):
- Dar AlUloom University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
will be made available to researchers upon reasonable request, in order to support further research and meta-analyses.
  Data to be Shared:
  Demographic data (e.g., age, gender)
  Baseline clinical characteristics
  Treatment allocation (coded)
  Outcome measures (e.g., clinical response, pain scores, lesion size)
  Adverse events and safety data
  Follow-up assessments
  Supporting Documents:
  Study protocol
  Statistical analysis plan
  Informed consent form (redacted)
  Case report forms (CRFs)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available beginning 6 months following publication and for up to 5 years. Data will be shared through secure data repositories or direct communication with the corresponding author, after review and approval of a formal data request, including a data use agreement.
Access Criteria: Access to IPD will be granted to qualified researchers affiliated with academic institutions, healthcare organizations, or non-profit research entities. Requests must include:
  A research proposal with clear scientific objectives and methods
  Evidence of ethical approval (if applicable)
  A signed data use agreement ensuring confidentiality, data protection, and responsible data handling
  Agreement not to attempt to re-identify individual participants
  Requests will be evaluated by the study team based on scientific merit, ethical considerations, and alignment with the purpose of the original study.